CLINICAL TRIAL: NCT04580225
Title: Randomized Comparison of PARtial Wrist Fusion With or Without Triquetral Excision (PARTE)
Acronym: PARTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Arthritis Society Canada (Unknown); Wrist Evaluation Canada (WECAN) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00099049
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Wrist Arthritis; Wrist Arthropathy; Scapholunate Advanced Collapse; Scaphoid Nonunion; Post-traumatic; Arthrosis; Arthritis; Musculoskeletal Diseases; Joint Diseases
Keywords: Post-traumatic wrist arthritis; Partial wrist fusions; Scapholunate advanced collapse; SLAC wrist; Scaphoid nonunion advanced collapse; SNAC wrist; Four-corner fusion; Bicolumnar wrist fusion; Three-corner fusion; Capitolunate fusion
MeSH Terms: conditions — Osteoarthritis; Arthritis; Musculoskeletal Diseases; Joint Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Partial Wrist Arthrodesis without Triquetral Excision (Active Comparator): Four-Corner Arthrodesis
  Interventions: Procedure: Four-Corner Arthrodesis
- Group B: Partial Wrist Arthrodesis with Triquetral Excision (Active Comparator): Three-Corner or Capitolunate Arthrodesis with Triquetral Excision
  Interventions: Procedure: Three-Corner or Capitolunate Arthrodesis with Triquetral Excision

INTERVENTIONS:
Procedure: Four-Corner Arthrodesis — Participants in Group A will receive a four-corner arthrodesis (fusion of the capitate, hamate, lunate, and triquetrum) with excision of the scaphoid.
  Arms: Group A: Partial Wrist Arthrodesis without Triquetral Excision
Procedure: Three-Corner or Capitolunate Arthrodesis with Triquetral Excision — Participants in Group B will receive a three-corner arthrodesis (fusion of the capitate, hamate, and lunate) or capitolunate arthrodesis (fusion of the capitate and lunate) with excision of the scaphoid and triquetrum.
  Arms: Group B: Partial Wrist Arthrodesis with Triquetral Excision

SUMMARY:
This randomized clinical trial (RCT) aims to compare clinical and radiographic outcomes of different partial wrist fusion techniques in participants with post-traumatic wrist arthritis. Participants with stage II or III scapholunate advanced collapse (SLAC) or scaphoid nonunion advanced collapse (SNAC) who meet the eligibility criteria will be randomly assigned to one of two parallel groups: Group A (partial wrist arthrodesis without triquetral excision i.e. four-corner arthrodesis), or Group B (partial wrist arthrodesis with triquetral excision i.e. three-corner or capitolunate arthrodesis with triquetral excision). The results of this study will provide evidence to guide surgeons in determining the ideal wrist fusion technique in the management of patients with post-traumatic wrist arthritis requiring surgery.

DETAILED DESCRIPTION:
This study has been designed as a multi-center double-blind prospective randomized clinical trial. Eligible participants will be adults presenting with SNAC or SLAC wrist arthritis who have been deemed an operative candidate and qualify for one of the following salvage techniques: four-corner arthrodesis (without triquetral excision) or three-corner/capitolunate arthrodeses with triquetral excision.

Once eligibility is confirmed, participants will be randomly assigned to one of two treatment arms. Participants in Group A will undergo four-corner arthrodesis; the scaphoid will be excised and the lunate, capitate, triquetrum, and hamate will be prepared and fused. Participants in Group B will undergo partial wrist arthrodesis with triquetral excision; the scaphoid and triquetrum will be excised. In the three-corner arthrodesis procedure, the articular surfaces between the lunate, capitate, and hamate will be prepared and fused. In the capitolunate arthrodesis procedure, only the articular surface between the lunate and capitate will be prepared and fused.

Eligible and consented participants will undergo a pre-operative study assessment and follow-up assessments at 6-weeks, 3-, 6-, and 12-months post-operative. Assessments will be conducted by an assessor blinded to participant treatment allocation. At each assessment, grip strength, wrist range of motion (ROM), Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire, Patient-Rated Wrist Evaluation (PRWE) questionnaire, and Visual Analog Scale (VAS) for pain will be completed. The work and sports/performing arts modules of the Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH), and the WOrk-Related Questionnaire for UPper extremity disorders (WORQ-UP), will be completed at baseline (pre-surgery) and at 12-months. Standard posteroanterior and lateral radiographs will be completed at all visits. Complications will be documented at each visit.

The primary outcome, grip strength, will be measured with a handheld dynamometer. Absolute values and percentage of their contralateral side will be compared between the two groups.

Statistical analysis will use the intention-to-treat approach with all outcomes attributed to the assigned group. Descriptive statistics will be used for group comparisons with independent t-tests for continuous and Pearson Chi-square or Fisher's Exact tests for categorical variables at baseline and for possible complications/adverse events. Linear Mixed Modeling (LMM), adjusted for age and sex, will compare outcomes between groups over the 12-month evaluation period. The level of significance will be set at α=0.05.

This study hypothesizes that partial wrist fusion with triquetral excision will lead to improved grip strength and ROM compared to four-corner arthrodesis. Considering the importance of ROM and grip strength in many activities of daily living and manual work, it is hypothesized that the group with triquetral excision (Group B) will have better patient-reported outcomes. We hypothesize no significant difference between the groups with regards to radiographic outcomes and complications.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a stage II or III scapholunate advanced collapse (SLAC) or scaphoid nonunion advanced collapse (SNAC) wrist and is a surgical candidate for the included surgical interventions

Exclusion Criteria:

* Participant has been diagnosed with other forms of wrist arthritis other than SLAC or SNAC
* Participant has significant arthritis of the ipsilateral hand/finger joint(s), major joint trauma, previous major wrist surgery, infection or neuromuscular pathology affecting the function of the ipsilateral upper extremity or ability to make a fist
* Participant has a physical or mental health condition preventing completion of consent or questionnaires
* Participant does not speak/read/understand English
* Participant has no fixed address or means of contact
* Participant is unwilling to complete necessary follow-ups
* Surgeon concludes that eligible salvage techniques are not appropriate at the time of surgery (based on injury characteristics or concomitant wrist pathology)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Grip Strength | Completed at baseline (pre-surgery), 3-, 6-, 12-months post-surgery
  Peak grip strength will be assessed using a hand-held dynamometer. Grip strength will be compared between groups over the 12-month evaluation period.

SECONDARY OUTCOMES:
Wrist Range of Motion (ROM) | Baseline, 3-, 6-, 12-months post-surgery
  Active and passive wrist ROM will be assessed using a goniometer. ROM will be compared between groups over the 12-month evaluation period.
Patient-Reported Outcomes Measurement Information System® (PROMIS) | Baseline, 6-weeks, 3-, 6-, 12-months post-surgery
  PROMIS questionnaire will be used to assess self-reported physical function, upper extremity, pain interference, emotional distress. PROMIS scores will be compared between groups over the 12-month evaluation period.
Patient-Rated Wrist Evaluation (PRWE) Questionnaire | Baseline, 6-weeks, 3-, 6-, 12-months post-surgery
  Pain and function from 0-10 will be self-reported using the PRWE. PRWE scores will be compared between groups over the 12-month evaluation period.
Visual Analog Scale (VAS) Pain Score | Baseline, 6-weeks, 3-, 6-, 12-months post-surgery
  Pain will be self-reported using VAS where zero equals no pain and 10 represents the worst possible pain. VAS pain scores will be compared between groups over the 12-month evaluation period.
Complications | 6-weeks, 3-, 6-, 12-months post-surgery
  Complications including infection and nonunion will be compared between groups over the 12-month evaluation period.
Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH) questionnaire - work and sports/performing arts modules | Baseline, 12-months post-surgery
  The work and sports/performing arts modules of the QuickDASH will be collected to measure the extent that participants experience limitations in their work and recreational activities, as applicable. Scores will be compared between groups.
WOrk-Related Questionnaire for UPper extremity disorders (WORQ-UP) questionnaire | Baseline, 12-months post-surgery
  The WORQ-UP will be collected to measure the extent that participants experience limitations in their work, as applicable. Scores will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Peter Lougheed Centre, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Western Hand & Upper Limb Facility, Sturgeon Community Hospital, St. Albert, Alberta
  - Lawson Health Research Institute, London, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan